CLINICAL TRIAL: NCT02391857
Title: The Clinical Study for the Identifying the Effect of Early Gastric Decompression on Improvement of Circulation During Advanced Cardiopulmonary Resuscitation
Brief Title: Early Gastric Decompression During Advanced Cardiopulmonary Resuscitation (EGD_ACLS)
Acronym: EGD_ACLS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Sang O, Park, Assistant Professor, Konkuk University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EGD2015
Record Dates: First submitted 2015-03-09; First posted 2015-03-18 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Out-of-Hospital Cardiac Arrest
Keywords: cardiopulmonary resuscitation; Gastric emptying
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EGDgroup (Experimental): Intervention (gastric decompression by naso(oro)-gastric tube insertion) was performed
  Interventions: Procedure: Gastric decompression

INTERVENTIONS:
Procedure: Gastric decompression — Insertion the Naso(Oro)-gastric tube for early gastric decompression during CPR

SUMMARY:
This study aimed to identify the effect of early gastric decompression on the improvement of circulation in arrest patients during cardiopulmonary resuscitation at the clinical setting of emergency department.

DETAILED DESCRIPTION:
Subjects and setting : adult sudden cardiac arrest patients in out of hospital, and transported to emergency department for advanced resuscitation treatment Interventions: first step, establish the advanced airway, after then insertion the naso (or oro)-gastric tube during CPR Data collection: live observation and review the automatically recoding data Missing or failed data should be collected and descriped Study period and sample size: numbers of participants necessary to identify the effect of interventions; 12 months or lesser were anticipated Analysis: All collected data can be analysed by Statistical programs

ELIGIBILITY:
Inclusion Criteria:

* Out of cardiac arrest patients who was transported to the emergency department for advanced resuscitation care

Exclusion Criteria:

* Do not attempted
* Inevitable death cofirmed at Emergency department
* Early recovery of spontaneous circulation before the intervention or sufficient collections of outcome data
* data loss
* others

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2018-01-01 (Actual)

PRIMARY OUTCOMES:
Evidence of improvement of circulatuion during CPR by evalution of increased end tidal CO2 (ETCO2) durig CPR | Within 10-20 min of CPR

OTHER OUTCOMES:
Mean compression depth of Chest compression | Within 10-20 min of CPR
Mean compression rate of Chest compression | Within 10-20 min of CPR
proportions of corrected release of Chest compression | Within 10-20 min of CPR

CONTACTS AND LOCATIONS:
Overall Officials: Sang O Park, MD, Study Director — Department of Emergency Medicine, School of medicine, Konkuk University
Locations (1):
- Department of Emergency Medicine, Konkuk University Medical center, Seoul, South Korea

REFERENCES:
- [Background] Wenzel V, Idris AH, Banner MJ, Kubilis PS, Band R, Williams JL Jr, Lindner KH. Respiratory system compliance decreases after cardiopulmonary resuscitation and stomach inflation: impact of large and small tidal volumes on calculated peak airway pressure. Resuscitation. 1998 Aug;38(2):113-8. doi: 10.1016/s0300-9572(98)00095-1. PMID 9863573
- [Background] Gabrielli A, Wenzel V, Layon AJ, von Goedecke A, Verne NG, Idris AH. Lower esophageal sphincter pressure measurement during cardiac arrest in humans: potential implications for ventilation of the unprotected airway. Anesthesiology. 2005 Oct;103(4):897-9. doi: 10.1097/00000542-200510000-00031. No abstract available. PMID 16192785
- [Background] Berg RA, Hemphill R, Abella BS, Aufderheide TP, Cave DM, Hazinski MF, Lerner EB, Rea TD, Sayre MR, Swor RA. Part 5: adult basic life support: 2010 American Heart Association Guidelines for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2010 Nov 2;122(18 Suppl 3):S685-705. doi: 10.1161/CIRCULATIONAHA.110.970939. PMID 20956221
- [Background] Wenzel V, Idris AH, Banner MJ, Kubilis PS, Williams JL Jr. Influence of tidal volume on the distribution of gas between the lungs and stomach in the nonintubated patient receiving positive-pressure ventilation. Crit Care Med. 1998 Feb;26(2):364-8. doi: 10.1097/00003246-199802000-00042. PMID 9468177
- [Background] von Goedecke A, Wagner-Berger HG, Stadlbauer KH, Krismer AC, Jakubaszko J, Bratschke C, Wenzel V, Keller C. Effects of decreasing peak flow rate on stomach inflation during bag-valve-mask ventilation. Resuscitation. 2004 Nov;63(2):131-6. doi: 10.1016/j.resuscitation.2004.04.012. PMID 15531063
- [Background] Aufderheide TP, Sigurdsson G, Pirrallo RG, Yannopoulos D, McKnite S, von Briesen C, Sparks CW, Conrad CJ, Provo TA, Lurie KG. Hyperventilation-induced hypotension during cardiopulmonary resuscitation. Circulation. 2004 Apr 27;109(16):1960-5. doi: 10.1161/01.CIR.0000126594.79136.61. Epub 2004 Apr 5. PMID 15066941